CLINICAL TRIAL: NCT04971902
Title: Pharmacist-led Pharmacogenomic Clinical Service Within the Program of All-inclusive Care for the Elderly (PACE)
Brief Title: Pharmacist-led Pharmacogenomic Clinical Service Within the Program of All-inclusive Care for the Elderly
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Tabula Rasa HealthCare (Industry)
Responsible Party: Sponsor
Other Study IDs: PGX-PACE-2020-001
Record Dates: First submitted 2021-02-15; First posted 2021-07-22 (Actual); Last update posted 2022-09-02 (Actual); Status verified 2022-09

CONDITIONS: Pharmacogenetic Testing; Elderly; Opioid Use; Pain; Pain, Acute; Pain, Chronic
MeSH Terms: conditions — Pain; Acute Pain; Chronic Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Pharmacogenetic Test — Cheek swab sample with PGx results lab analysis

SUMMARY:
Pharmacist-led pharmacogenomics (PGx) clinical services and medication safety reviews are currently being offered to PACE organizations under the direction of licensed healthcare prescribers by CareKinesis d/b/a Tabula Rasa HealthCare. This project aims to include patients enrolled in PACE organizations with chronic pain and who are prescribed CYP2D6 activated opioids. PGx testing will be performed by contractual PGx vendor with TRHC. PGx results will be integrated into TRHC's proprietary Clinical Decision Support System (Medication Risk Mitigation™ Matrix, CareKinesis, Moorestown, NJ) that guides pharmacists to identify drug-drug interactions (DDIs), drug-gene interactions (DGIs), and drug-drug-gene interactions (DDGIs).16 Clinical pharmacists will translate PGx results combined with a comprehensive DDI review into actionable clinical decisions. Clinical pharmacists will provide medication therapy management recommendation to address medication problems to the PACE prescriber (physician). PACE prescribers will review the pharmacist's recommendation, and based on their clinical assessment, the prescriber will decide whether or not to implement the opioid therapy recommendation.

DETAILED DESCRIPTION:
Tabula Rasa HealthCare (TRHC), doing business as CareKinesis, is the first national pharmacy that provides science-based medication risk identification and mitigation technologies and services. CareKinesis utilizes medication decision support tools and pharmacists certified in geriatrics to provide pharmacy services for various healthcare organizations including PACE organizations.

Program of All-inclusive Care for the Elderly (PACE) is a Medicare-Medicaid program that provides comprehensive medical and supportive services to individuals >55 years of age who are certified by their state as needing nursing home care. As an alternative to institutionalization, PACE helps these individuals live safely in their community. The aim of PACE is to improve overall quality of life in four domains (physical, psychological, social, and spiritual) using a multidisciplinary approach. In the United States, the vast majority of PACE organizations collaborate with one pharmacy to dispense drugs, in addition to other pharmacy services, for their population of participants.15 Presently, CareKinesis services more than 35 PACE organizations, including approximately 75 PACE sites, across the country. As a national PACE pharmacy provider since 2011, CareKinesis focuses on improving medication regimens to reduce medication-related risks while enhancing economic, clinical and humanistic outcomes.

Study Design Pharmacist-led pharmacogenomics (PGx) clinical services and medication safety reviews are currently being offered to PACE organizations under the direction of licensed healthcare prescribers by CareKinesis d/b/a Tabula Rasa HealthCare. This project aims to include patients enrolled in PACE organizations with chronic pain and who are prescribed CYP2D6 activated opioids. PGx testing will be performed by a contractual PGx vendor with TRHC. PGx results will be integrated into TRHC's proprietary Clinical Decision Support System (Medication Risk Mitigation™ Matrix, CareKinesis, Moorestown, NJ) that guides pharmacists to identify drug-drug interactions (DDIs), drug-gene interactions (DGIs), and drug-drug-gene interactions (DDGIs).16 Clinical pharmacists will translate PGx results combined with a comprehensive DDI review into actionable clinical decisions. Clinical pharmacists will provide medication therapy management recommendation to address medication problems to the PACE prescriber (physician). PACE prescribers will review the pharmacist's recommendation, and based on their clinical assessment, the prescriber will decide whether or not to implement the opioid therapy recommendation.

The measurement of health-related quality of life (QoL) and pain assessment using the EQ-5D survey, and numerical rating scale (NRS) for pain will be performed during the study by PACE prescribers or the PACE interdisciplinary team (IDT) as follows:

* Health-related quality of life questionnaire (EQ-5D) will be performed at baseline and at the completion of the study (visits 1 and 3, respectively)
* NRS for pain will be performed at baseline (before the PGx testing), 1-2 and 2-3 weeks after TRHC's pharmacist recommendations (visits 1, 2 and 3, respectively) All PACE patients will continue to receive usual medical care throughout the study. Changes to drug regimens will be at the discretion of the patients' PACE prescribers.

ELIGIBILITY:
Inclusion Criteria:

1. Patient enrolled in a PACE organization during the implementation period; and,
2. PACE organization contractually receiving pharmacy services from CareKinesis
3. Patient prescribed a CYP2D6 activated opioid, namely codeine, hydrocodone, oxycodone and/or tramadol
4. Patients with chronic non-cancer pain (CNCP)
5. Patient's prescriber orders a PGx test based upon his/her determination that the patient could potentially benefit from PGx testing
6. Patient is able to read, understand, and provide informed consent to participate

Exclusion Criteria:

1. Patient prescribed an opioid that is not metabolized by CYP2D6 including, but not limited to, oxymorphone, morphine, hydromorphone
2. Have taken an investigational product in the last 30 days
3. Current use of illicit substances
4. Immediate family members of site staff, or site staff may not be enrolled in the study without first obtaining IRB authorization
5. Any other medical, cognitive or physical abnormality, disease, or disorder that would prohibit the patient from completing study procedures in the judgement of the investigator

Min Age: 55 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Program of All-inclusive Care for the Elderly (PACE) is a Medicare-Medicaid program that provides comprehensive medical and supportive services to individuals >55 years of age who are certified by their state as needing nursing home care. As an alternative to institutionalization, PACE helps these individuals live safely in their community
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Measure the feasibility of Clinical Decision Support System (MedWise(TM)) for CYP2D6 opioid prescription and PGx recommendations by usability and acceptability through physician and pharmacist questionnaire. | 6 months
  Quantitative data reported via survey
Measure the feasibility of Clinical Decision Support System (MedWise(TM)) for PGx recommendations by acceptability through physician and pharmacist questionnaire. | 6 months
  Quantitative data reported via survey
Measure the feasibility of Clinical Decision Support System (MedWise(TM)) for PGx recommendations by usability through physician and pharmacist questionnaire. | 6 months
  Quantitative data reported via survey
Analyze patient medication information for PGx- and DDI-guided recommendations using MedWise(TM) a proprietary clinical decision support system by Tabula Rasa HealthCare. | 6 months
  Quantitative (software is proprietary and patented)
Analyze clinician uptake of PGx- and DDI-guided recommendations using MedWise(TM) a proprietary clinical decision support system by Tabula Rasa HealthCare. | 6 months
  Quantitative (software is proprietary and patented)
Validate patient QOL questionnaire for disease-related information | 6 months
  Quantitative data measured by percentage of improvement for DDI-guided recommendations based on PGx results
Validate patient QOL questionnaire for pharmacogenetics information | 6 months
  Quantitative data measured by percentage of improvement for DDI-guided recommendations based on PGx results
Validate patient QOL questionnaire for medication-related information, and pharmacogenetics information | 6 months
  Quantitative data measured by percentage of improvement for DDI-guided recommendations based on PGx results
Validate patient QOL questionnaire for socio-demographics | 6 months
  Quantitative data measured by percentage of improvement for DDI-guided recommendations based on PGx results

CONTACTS AND LOCATIONS:
Overall Officials: Veronique Michaud, PhD, Principal Investigator — Tabula Rasa HealthCare
Locations (1):
- Tabula Rasa HealthCare Precision Pharmacotherapy Research and Development Institute, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No